CLINICAL TRIAL: NCT02760485
Title: An Open-Label Phase 1/2 Study of Itacitinib (INCB039110) in Combination With Ibrutinib in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Itacitinib (INCB039110) in Combination With Ibrutinib in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-206
Record Dates: First submitted 2016-05-02; First posted 2016-05-03 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: Diffuse large B-cell lymphoma; Relapsed Diffuse large B-cell lymphoma; Refractory Diffuse large B-cell lymphoma; activated B cell; germinal center B-cell; non-Hodgkin lymphoma; JAK1 inhibitor; Bruton's tyrosine kinase (BTK) inhibitor
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — itacitinib; INCB039110; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- itacitinib + ibrutinib (Experimental)
  Interventions: Drug: itacitinib; Drug: ibrutinib

INTERVENTIONS:
Drug: itacitinib — Phase 1 will evaluate itacitinib at the protocol-specified starting dose, with a possible increase or decrease depending on tolerability. Phase 2 will evaluate the recommended dose determined in Phase 1.
  Other Names: INCB039110
Drug: ibrutinib

SUMMARY:
The purpose of this study is to evaluate the safety/tolerability and efficacy of itacitinib in combination with ibrutinib in subjects with relapsed or refractory diffuse large B-cell lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of DLBCL.

  * Phase 1: any DLBCL subtype.
  * Phase 2: activated B-cell or unclassifiable subtypes confirmed by immunohistochemistry using the Hans algorithm
* Relapsed or refractory DLBCL, defined as having received at least 1 but no more than 3 prior treatment regimens and ineligible for high-dose chemotherapy/autologous stem cell transplant.
* Fluorodeoxyglucose-avid disease (based on local evaluation) per the Lugano Classification. Fluorodeoxyglucose-avid disease is defined as disease with a 5-point scale score of 4 or 5.
* Archived tumor tissue (block or 15-20 unstained slides) available, or be willing to undergo an incisional or excisional lymph node biopsy of accessible adenopathy (or, in less accessible lymph nodes, 4 to 8 core biopsies).
* At least 1 measurable (≥ 2 cm in longest dimension) lesion on CT scan or magnetic resonance imaging (MRI).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

Exclusion Criteria:

* Transformed DLBCL or DLBCL with coexistent histologies (eg, follicular or mucosa-associated lymphoid tissue lymphoma).
* Primary mediastinal (thymic) large B-cell lymphoma.
* Known central nervous system lymphoma (either primary or metastatic).
* Allogeneic stem cell transplant within the previous 6 months, or active graft versus host disease following allogeneic transplant.
* Use of immunosuppressive therapy within 28 days of starting study treatment. Immunosuppressive therapy includes but is not limited to cyclosporine A, tacrolimus, or high-dose corticosteroids. Subjects receiving corticosteroids must be at a dose level ≤ 10 mg/day within 7 days of initiating study treatment.
* Prior or concurrent therapy with a Janus kinase inhibitor or Bruton's tyrosine kinase inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — Incyte Corporation
Locations (21):
- United States (21):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Pacific Shores Medical Group, Long Beach, California
  - LAC-USC Medical Center/Kenneth Norris Jr Cancer Hospital, Los Angeles, California
  - Moores UC San Diego Cancer Center, San Diego, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Georgia Regents Research Institute, Augusta, Georgia
  - University of Maryland Cancer Center, Baltimore, Maryland
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Michigan State University Breslin Cancer Center, Lansing, Michigan
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Regional Cancer Center Associates, LLC, Little Silver, New Jersey
  - Roswell Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Toledo Clinic Cancer Centers, Toledo, Ohio
  - Tulsa Cancer Center, Tulsa, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Houston Methodist Cancer Center, Houston, Texas
  - Northwest Medical Specialists & Research Institute, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 12 study centers in the United States.
Groups:
- Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD: Participants received oral itacitinib 300 milligrams (mg) once daily (QD) plus oral ibrutinib 560 mg QD until treatment discontinuation criteria were met.
- Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD; Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD: Participants received oral itacitinib 400 mg QD plus oral ibrutinib 560 mg QD until treatment discontinuation criteria were met.
Period: Phase 1
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Started | 7 | 7 | 0
Completed | 0 | 0 | 0
Not Completed | 7 | 7 | 0
Not completed — Death | 3 | 6 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Amendment Removed Survival Follow-up | 0 | 1 | 0
Not completed — Unknown; Did Not Complete End-of-Study Visit | 1 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Started | 0 | 0 | 19
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 19
Not completed — Death | 0 | 0 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Progressive Disease | 0 | 0 | 1
Not completed — Unknown; Did Not Complete End-of-Study Visit | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: In Phase 1, Baseline data were collected for members of the Safety Run-In Population, defined as all participants enrolled in the Phase 1 portion of the study who received at least 1 dose of study drug. In Phase 2, Baseline data were collected for members of the Intent-to-Treat Population, defined as all participants enrolled in the Phase 2 portion of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Total
Number analyzed (Participants) | 6 | 7 | 19 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (10.42) | 67.0 (13.39) | 72.1 (14.25) | 70.6 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 6 | 13
  Male | 4 | 2 | 13 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 6 | 4 | 13 | 23
  Black/African-American | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 2
  Captured as "Other" | 0 | 1 | 3 | 4
  Missing | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 4 | 3 | 13 | 20
  Not Reported | 1 | 0 | 3 | 4
  Unknown | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and until 30 days after the last dose of study drug.
Time Frame: up to 285 days
Population: Safety Run-In Population: all participants enrolled in the Phase 1 portion of the study who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 6 | 7 | 0
Participants | 6 | 7 |

2. Primary Outcome: Phase 1: Number of Participants With Any Grade 3 or Higher TEAE
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and until 30 days after the last dose of study drug. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated.
Time Frame: up to 285 days
Population: Safety Run-In Population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 6 | 7 | 0
Participants | 5 | 5 |

3. Primary Outcome: Phase 1: Number of Participants With Any Dose-limiting Toxicity (DLT)
Description: A DLT was defined as the occurrence of any protocol-defined toxicities occurring up to and including Study Day 28, except those with a clear alternative explanation (e.g., disease progression) or transient (≤72 hours) abnormal laboratory values without associated clinically significant signs or symptoms based on investigator determination. All DLTs were assessed by the investigator using Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria. In order to be included in the tolerability review, subjects must have received the cohort-specific dose of INCB039110 and ibrutinib for at least 75% of the days during the 28-day surveillance period or have experienced a DLT.
Time Frame: up to Day 28
Population: Safety Run-In Population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 6 | 7 | 0
Participants | 0 | 1 |

4. Primary Outcome: Phase 2: Objective Response Rate (ORR), Defined as the Percentage of Participants Achieving Either a Complete Response (CR) or a Partial Response (PR), Per the Modified Lugano Classification for Diffuse Large B-cell Lymphoma (DLBCL)
Description: CR: (1) target nodes/nodal masses of lymph nodes/extralymphatic sites regressed to ≤1.5 centimeters (cm) in the longest dimension transverse diameter of lesion (LDi); (2) absence of non-measured lesions; (3) organ enlargement regressed to normal; (4) no new lesions; (5) normal bone marrow morphology; if indeterminate, immunohistochemistry negative. PR: (1) lymph nodes/extralymphatic sites: ≥50% decrease in the sum of the product of perpendicular diameters for multiple lesions of up to 6 target measurable nodes/extranodal sites; if lesion is too small to measure on computed tomography, assign 5 millimeters (mm) × 5 mm as default; if no longer visible, 0 mm × 0 mm. For node >5 mm × 5 mm but smaller than normal, use actual measurement; (2) absent/regressed non-measured lesions, no increase; (3) organ enlargement; spleen regressed by >50% in length beyond normal; (4) no new lesions.
Time Frame: up to 1538 days
Population: Intent-to-Treat (ITT) Population: all participants enrolled in the Phase 2 portion of the study. The confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 0 | 0 | 19
percentage of participants |  |  | 26.3 [10.99 to 47.58]

5. Secondary Outcome: Phase 1: ORR, Defined as the Percentage of Participants Achieving Either a CR or a PR, Per the Modified Lugano Classification for DLBCL
Description: CR: (1) target nodes/nodal masses of lymph nodes/extralymphatic sites regressed to ≤1.5 cm in the LDi; (2) absence of non-measured lesions; (3) organ enlargement regressed to normal; (4) no new lesions; (5) normal bone marrow morphology; if indeterminate, immunohistochemistry negative. PR: (1) lymph nodes/extralymphatic sites: ≥50% decrease in the sum of the product of perpendicular diameters for multiple lesions of up to 6 target measurable nodes/extranodal sites; if lesion is too small to measure on computed tomography, assign 5 mm × 5 mm as default; if no longer visible, 0 mm × 0 mm. For node >5 mm × 5 mm but smaller than normal, use actual measurement; (2) absent/regressed non-measured lesions, no increase; (3) organ enlargement; spleen regressed by >50% in length beyond normal; (4) no new lesions.
Time Frame: up to 250 days
Population: Safety Run-in Population. The confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 6 | 7 | 0
percentage of participants | 33.3 [6.28 to 72.87] | 57.1 [22.53 to 87.12] |

6. Secondary Outcome: Phase 2: Duration of Response (DOR): Time From the First Overall Response Contributing to an Objective Response (CR or PR) to the Earlier of the Participant's Death and the First Overall Response of Progressive Disease, Per the Lugano Classification
Description: Disease progression requires ≥1 of the following: (1) an abnormal individual node/lesion with all of the following: (a) LDi > 1.5 cm; (b) increase by ≥50% from cross product of the LDi and the perpendicular diameter (PPD) nadir; (c) increase in LDi or the shortest axis perpendicular to the LDi (SDi) from nadir: (i) 0.5 cm for lesions ≤2 cm; (ii) 1.0 cm for lesions > 2 cm. (2) For splenomegaly, the splenic length must increased by 50% of the extent of its prior increase beyond baseline. If no prior splenomegaly, must increase by at least 2 cm from baseline. (3) New/recurrent splenomegaly. (4) New/clear progression of preexisting nonmeasured lesions. (5) Regrowth of previously resolved lesions. (6) A new node > 1.5 cm in any axis. (7) A new extranodal site > 1.0 cm in any axis; if < 1.0 cm in any axis, its presence must be unequivocal/attributable to lymphoma. (8) Assessable disease of any size unequivocally attributable to lymphoma. (9) New or recurrent involvement of the bone marrow.
Time Frame: up to 947 days
Population: ITT Population. Participants who achieved a CR or a PR per Lugano Classification for DLBCL were analyzed. The 90% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 0 | 0 | 5
months |  |  | 8.80 [1.94 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died.

7. Secondary Outcome: Phase 2: Durable Response Rate (DRR)
Description: DRR=percentage of participants with a CR or PR, per Lugano Classification, for ≥16 weeks since the time from the first overall response contributing to an objective response (CR or PR). CR: (1) target nodes/nodal masses of lymph nodes/extralymphatic sites regressed to ≤1.5 cm in the LDi; (2) absence of non-measured lesions; (3) organ enlargement regressed to normal; (4) no new lesions; (5) normal bone marrow morphology; if indeterminate, immunohistochemistry negative. PR: (1) lymph nodes/extralymphatic sites: ≥50% decrease in the sum of the product of perpendicular diameters for multiple lesions of up to 6 target measurable nodes/extranodal sites; if lesion is too small to measure on computed tomography, assign 5 mm × 5 mm as default; if no longer visible, 0 mm × 0 mm. For node >5 mm × 5 mm but smaller than normal, use actual measurement; (2) absent/regressed non-measured lesions, no increase; (3) organ enlargement; spleen regressed by >50% in length beyond normal; (4) no new lesions.
Time Frame: up to 1538 days
Population: ITT Population. Participants who achieved a CR or a PR per Lugano Classification were analyzed. The confidence interval was calculated based on the exact method for binomial distribution.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 0 | 0 | 5
percentage of participants |  |  | 60.0 [18.93 to 92.36]

8. Secondary Outcome: Phase 2: Progression-free Survival (PFS), Defined as the Time From the First Dose to the Earlier Date of Death Due to Any Cause or Disease Progression Determined by Objective Radiographic Disease Assessments
Description: as for outcome 6
Time Frame: up to 1538 days
Population: ITT Population. The 90% confidence interval was calculated using the Brookmeyer and Crowley's method.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 0 | 0 | 19
months |  |  | 3.17 [1.38 to 7.10]

9. Secondary Outcome: Phase 2: Number of Participants With Any TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and until 30 days after the last dose of study drug.
Time Frame: up to 1573 days
Population: Safety Evaluable Population: all participants enrolled in the Phase 2 portion of the study who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 0 | 0 | 19
Participants |  |  | 19

10. Secondary Outcome: Phase 2: Number of Participants With Any Grade 3 or Higher TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug and until 30 days after the last dose of study drug. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4: life-threatening consequences; urgent intervention indicated.
Time Frame: up to 1573 days
Population: Safety Evaluable Population
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phase 1; Cohort 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Phase 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD
Number analyzed (Participants) | 0 | 0 | 19
Participants |  |  | 16

ADVERSE EVENTS:
Time Frame: Phase 1 participants were monitored for up to 285 days. Phase 2 participants were monitored for up to 1573 days.
Description: Treatment-emergent adverse events (AEs reported for the first time or the worsening of pre-existing AEs after the first dose and until 30 days after the last dose of study drug) are reported for members of the Phase 1 Safety Run-In Population and the Phase 2 Safety Evaluable Population (all enrolled participants who received ≥1 dose of study drug).
Groups:
- Phases 1 and 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD: Participants in Cohort 2 of Phase 1 and in Phase 2 received oral itacitinib 400 mg QD plus oral ibrutinib 560 mg QD until treatment discontinuation criteria were met.
- Total: Total
Arm/Group | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD | Phases 1 and 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD | Total
All-Cause Mortality (participants affected / at risk) | 2/6 | 19/26 | 21/32
Serious Adverse Events (participants affected / at risk) | 4/6 | 18/26 | 22/32
Other Adverse Events (participants affected / at risk) | 6/6 | 26/26 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD (N=6) | Phases 1 and 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD (N=26) | Total (N=32)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 4 (4) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (4) | 3 (4)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1; Cohort 1: Itacitinib 300 mg QD + Ibrutinib 560 mg QD (N=6) | Phases 1 and 2: Itacitinib 400 mg QD + Ibrutinib 560 mg QD (N=26) | Total (N=32)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 7 (7) | 9 (9)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 3 (3)
Asthenia (General disorders) | 2 (2) | 2 (2) | 4 (4)
Blood cholesterol increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 2 (4) | 2 (4)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (3) | 9 (9) | 11 (12)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 7 (8) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 9 (10) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 9 (14) | 11 (16)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 7 (7) | 8 (8)
Dizziness postural (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (8) | 8 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 4 (6)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 4 (5)
Fatigue (General disorders) | 3 (3) | 12 (15) | 15 (18)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (4) | 3 (3) | 4 (7)
Hypertension (Vascular disorders) | 1 (3) | 3 (3) | 4 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 4 (4)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (10) | 9 (12)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 2 (3)
Oedema peripheral (General disorders) | 0 (0) | 4 (5) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 4 (7) | 4 (7)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 6 (6) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Tongue eruption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 3 (4)
Vision blurred (Eye disorders) | 1 (1) | 3 (3) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Wound infection pseudomonas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT02760485/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT02760485/SAP_001.pdf